CLINICAL TRIAL: NCT01499667
Title: A 32-week, Patient- and Rater-blinded, Randomized, Multi-center, Parallel-group Study to Evaluate Disease Control and Safety in Patients With Relapsing Remitting Multiple Sclerosis Transferred From Previous Treatment With Natalizumab to Fingolimod (FTY720)
Brief Title: Disease Control and Safety in Patients With Relapsing Remitting Multiple Sclerosis (RRMS) Switching From Natalizumab to Fingolimod
Acronym: TOFIINGO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on recent publications, determination of natalizumub washout period was no longer relevant.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2324; 2011-001442-15 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-12-26 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: Relapsing remitting multiple sclerosis; multiple sclerosis (MS); safety; tolerability; health outcomes; fingolimod; disease control; MRI
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 8-week washout + Fingolimod (FTY720) (Experimental): 8-week washout (8 weeks no treatment) followed by 24 weeks of treatment with fingolimod 0.5mg once a day
  Interventions: Drug: Fingolimod
- 12-week washout + Fingolimod (FTY720) (Experimental): 12-week washout (8 weeks no treatment and 4 weeks placebo) followed by 20 weeks of treatment with fingolimod 0.5mg once a day
  Interventions: Drug: Fingolimod; Drug: Placebo
- 16-week washout + Fingolimod (FTY720) (Experimental): 16-week washout (8 weeks no treatment and 8 weeks placebo) followed by 16 weeks of treatment with fingolimod 0.5mg once a day
  Interventions: Drug: Fingolimod; Drug: Placebo

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5 mg capsules for oral administration once daily
Drug: Placebo — Matching placebo in capsules for oral administration once daily.
  Arms: 12-week washout + Fingolimod (FTY720); 16-week washout + Fingolimod (FTY720)

SUMMARY:
This study evaluated disease control during different lengths of treatment transition from natalizumab to fingolimod.

DETAILED DESCRIPTION:
Patient were screened, signed an informed consent at visit 1, at the 2nd visit, all patient received a baseline infusion of Natalizumub and subsequently randomized to one of 3 treatment arms. At the randomization visit, the Washout Phase started, and eligible patients were randomized 1:1:1 to one of three treatment groups:

* 8-week washout (8 weeks no treatment) followed by 24 weeks of treatment with fingolimod,
* 12-week washout (8 weeks no treatment and 4 weeks placebo) followed by 20 weeks of treatment with fingolimod, or
* 16-week washout (8 weeks no treatment and 8 weeks placebo) followed by 16 weeks of treatment with fingolimod.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* Have relapsing remitting multiple sclerosis
* Have been on treatment with natalizumab for at least 6 months prior to screening and discontinuation is an option.

Exclusion Criteria:

Patients with:

* History of chronic immune disease
* Crohn's disease
* Certain cancers
* Uncontrolled diabetes
* Certain eye disorders
* Negative for varicella-zoster virus IgG antibodies
* Certain hepatic conditions
* Low white blood cell count
* On certain immunosuppressive medications or heart medications
* Resting heart rate less than 45 bpm.
* Certain heart conditions or certain lung conditions
* Inability to undergo MRI scans

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- Australia (2):
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
- Novartis Investigative Site, Vienna, Austria
- Czechia (2):
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Novartis Investigative Site, Helsinki, Finland
- Germany (19):
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Celle, Germany
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Kandel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neuburg am Inn
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Budapest, Hungary
- Israel (2):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Cefalù, PA
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Basel, Switzerland

REFERENCES:
- [Derived] Derfuss T, Kovarik JM, Kappos L, Savelieva M, Chhabra R, Thakur A, Zhang Y, Wiendl H, Tomic D. alpha4-integrin receptor desaturation and disease activity return after natalizumab cessation. Neurol Neuroimmunol Neuroinflamm. 2017 Aug 25;4(5):e388. doi: 10.1212/NXI.0000000000000388. eCollection 2017 Sep. PMID 28856176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 158 patients screened, 142 patients were randomized.
Pre-assignment Details: 142 Participants were randomized to 3 washout groups in a ratio of 1:1:1
Period: Overall Study
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Started | 50 (Started" indicates randomized as well as safety population.) | 42 | 50
Full Analysis Set (FAS) | 49 (One randomized patient did not receive natalizumub at screening, which was a requirement for FAS.) | 42 | 50
Modified Full Analysis Set | 41 (mFAS included all FAS patients who completed 8 wks of fingolimod treatment with MRI scan) | 29 | 39
Completed | 41 | 31 | 40
Not Completed | 9 | 11 | 10
Not completed — administrative problems | 4 | 5 | 5
Not completed — Protocol Violation | 1 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set includes all subjects who receive a randomization number, regardless of whether or not they receive study medication.
Groups:
- 16-week Washout + Fingolimod (FTY720): 16-week washout (8 weeks no treatment and 8 weeks placebo) followed by 16 weeks of treatment with fingolimod
- Total: Total of all reporting groups
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720) | Total
Number analyzed (Participants) | 50 | 42 | 50 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (10.102) | 41.9 (7.445) | 41.8 (8.552) | 41.6 (8.780)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 21 | 32 | 92
  Male | 11 | 21 | 18 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Active (New or Newly Enlarging) T2 Lesions From the Last Natalizumab Infusion (Baseline) Through 8 Weeks of Fingolimod Treatment
Description: Active lesions were measured on brain MRI scans, performed at week 8, compared to the prior scan. The primary variable was analyzed by fitting a negative binomial regression model adjusted for washout group.
Time Frame: Number of active T2 lesions from last natalizumab dose through 8 weeks of fingolimod treatment
Population: The modified Full Analysis Set (mFAS) included all patients in the Full Analysis Set who completed 8 weeks of fingolimod treatment and provided an MRI scan at this time point. The analysis of primary variable was performed on the mFAS.
Measure: Mean (Standard Deviation); unit: Count of Active T2 Lesions
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 41 | 29 | 39
Count of Active T2 Lesions | 2.1 (7.24) | 1.7 (3.78) | 8.2 (16.81)

2. Secondary Outcome: Number of Active (New or Newly Enlarging) T2 Lesions From the Last Natalizumab Infusion (Baseline) up to the Initiation of Fingolimod Treatment
Description: Lesions were measured by MRIs and the number of active (new or newly enlarging) T2 lesions was calculated from baseline to beginning of treatment.
Time Frame: 8, 12 and 16 weeks (number of active T2 lesions during the washout period only)
Population: The Full Analysis Set (FAS) included all randomized patients who had at least one recorded dose of natalizumab at the Week 0 visit, analyzed according to the washout group assigned at randomization
Measure: Mean (Standard Deviation); unit: Count of active T2 lesions
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 49 | 42 | 50
Count of active T2 lesions | 0.4 (2.71) | 2.1 (11.15) | 3.6 (7.54)

3. Secondary Outcome: Number of Active (New or Newly Enlarging) T2 Lesions During the First 8 Weeks of Fingolimod Treatment
Description: Lesions were measured by MRIs and the number of active (new or newly enlarging) T2 lesions was calculated for first 8 weeks of fingolimod treatment.
Time Frame: Number of active T2 lesions during 8 wks of fingolimod treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Count of Active T2 Lesions
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 49 | 42 | 50
Count of Active T2 Lesions | 1.5 (4.56) | 2.1 (5.50) | 4.2 (10.24)

4. Secondary Outcome: Number of Active (New or Newly Enlarging) T2 Lesions During the 24 Weeks After the Last Natalizumab Infusion (Baseline)
Description: Lesions will be measured by MRIs and the number of active (new or newly enlarging) T2 lesions will be calculated for 24 weeks from baseline.
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Count of Active T2 Lesions
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 49 | 42 | 50
Count of Active T2 Lesions | 3.2 (10.07) | 4.4 (16.01) | 7.7 (16.28)

5. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) by Washout Group
Description: Kurtzke's Expanded Disability Status Scale (EDSS) measures the changes in neurologic impairment, either chronic (progression over time), or acute (MS relapses). The EDSS steps range from 0 (normal) to 10 (death due to MS). Relapse severity is assessed based on severity of neurologic impairment as evaluated using the EDSS.
Time Frame: Baseline to week 16 and week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 49 | 42 | 50
Units on a scale
  Week 16 (n=40, 33, 39) | 0.11 (0.330) | -0.03 (0.529) | 0.23 (0.706)
  Week 32 (n= 40,30,39) | 0.11 (0.625) | -0.13 (0.524) | 0.08 (0.748)

6. Secondary Outcome: Cumulative Number of Gadolinium-enhancing T1 Lesions From the Last Natalizumab Infusion
Description: Gadolinium-enhancing lesions will be measured on post-contrast T1-weighted brain MRI scans
Time Frame: 8 weeks and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of Gd enhanced T1 Lesions
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 49 | 42 | 50
Number of Gd enhanced T1 Lesions
  Week 8 (n=1,1,0) | 25.0 (0) | 2.0 (0) | NA (NA) — No data collected for this time point
  Week 24 (n=10,12,21) | 6.3 (9.45) | 3.4 (4.54) | 3.6 (4.49)

7. Secondary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE) and Death During Washout Period
Description: Adverse events were summarized by the number of patients having any adverse event overall.
Time Frame: Baseline to maximum of 16 weeks
Population: The Safety Set included all randomized patients, analyzed according to the washout group most closely corresponding to the day on which they first received fingolimod
Measure: Number; unit: participants
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 50 | 42 | 50
participants
  Any Adverse Events | 13 | 12 | 25
  Serious Adverse Events | 0 | 0 | 1
  Death | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE) and Death During Fingolimod Treatment
Description: Adverse events were summarized by the number of patients having any adverse event overall.
Time Frame: Baseline to maximum of 16 weeks
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Number analyzed (Participants) | 50 | 42 | 50
participants
  Any Adverse Events | 35 | 20 | 28
  Serious Adverse Events | 2 | 5 | 3
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety Set (SS): The Safety Set included all randomized patients, analyzed according to the washout group most closely corresponding to the day on which they first received fingolimod. Safety and tolerability analysis were performed on the SS unless otherwise specified.
Arm/Group | 8-week Washout + Fingolimod (FTY720) | 12-week Washout + Fingolimod (FTY720) | 16-week Washout + Fingolimod (FTY720)
Serious Adverse Events (participants affected / at risk) | 2/50 | 5/42 | 4/50
Other Adverse Events (participants affected / at risk) | 17/50 | 7/42 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 8-week Washout + Fingolimod (FTY720) (N=50) | 12-week Washout + Fingolimod (FTY720) (N=42) | 16-week Washout + Fingolimod (FTY720) (N=50)
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1
Heart rate decreased (Investigations) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 8-week Washout + Fingolimod (FTY720) (N=50) | 12-week Washout + Fingolimod (FTY720) (N=42) | 16-week Washout + Fingolimod (FTY720) (N=50)
Nasopharyngitis (Infections and infestations) | 7 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 3 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 3
Headache (Nervous system disorders) | 5 | 3 | 10
Depression (Psychiatric disorders) | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated due to new data on nataluzimab washout prior to treatment with other disease modifying treatments. The power to detect statistically significant differences between the washout groups based on the (-)binomial is estimated 30-40%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.